CLINICAL TRIAL: NCT06790992
Title: Relıabılıty and Valıdıty of the Supıne-to-stand Test As a Measure of Functional Motor Competence In People Wıth Multiple Sclerosis
Brief Title: Relıabılıty and Valıdıty of the Supıne-to-stand Test Wıth Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, Physiotherapy and Rehabilitation Department, Assistant Professor, Sanko University
Other Study IDs: SANKO University: 2024/6-01
Record Dates: First submitted 2024-11-07; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: Supine-to-Stand Test (SST) requires muscle strength, flexibility, and dynamic balance and can be used as a marker of functional motor competence in patients with Multiple Sclerosis (pwMS).

Objectives: To investigate the reliability and validity of SST in pwMS. Methods: Muscle strength was measured using digital goniometer for plantar and dorsiflexor in pwMS (n=44). Manual dexterity was assessed through the 9-hole Peg Test (9HPT). Balance was evaluated using with Berg Balance Test (BBT). Walking speed was assessed using Six-minute Walk test (6MWT). Timed up and go test (TUG), Activity-spesific Balance Confidence scale was used for fear of falling. Quality of life was assessed with MSQOL-54.

Results: The test's intraclass correlation was 0.984 (95% CI 0.801-0.995). Significant moderate correlations were found between SST and BBT (r=-0.547, p=0.001), TUG (r=0.619, p<0.001), and 6MWT (r=-0.642, p<0.001). A moderate correlation was also found between dominant side plantar flexor strength and SST (r=0.349, p=0.043), but not non-dominant side and bilaterally dorsi flexors (p>0.05). Additionally, no significant correlation was found between SST and bilaterally 9HPT, MSQOL-54 (p>0.05).

Conclusion: This study establishes SST as a reliable and valid tool for assessing functional motor competence in pwMS.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a demyelinating, inflammatory, neurodegenerative and progressive disease that causes varying degrees of disability in mobility and functional activities and affects social participation . Common symptoms in MS patients are usually; tone changes, loss of strength in the lower extremities, spasticity, balance and coordination problems, problems, falls, and walking problems . It becomes very difficult for patients with MS (pwMS) to transition between movements and positions considering these symptoms .

The ability to stand from a supine position is the basis for people's ability to get out of bed every day. This activity is very important in situations such as being able to stand by controlling movement while standing and getting up after falls . Supine-to-stand ability requires muscle strength, flexibility, and dynamic balance . The movement includes complex sub- sequential patterns such as sit-to-stand. Factors such as duration, quality of the subsections, and sitting balance also affect supine-to-stand ability . Besides, supine-to-stand ability is seen as indicator for establishing and maintaining bipedal independence. It is evaluated in the pediatric group as fundamental movement skills and motor competence in relation to functional capacity . Therefore, it is essential to determine the clinical applicability of the supine-to stand test (SST) for assessing the competence of pwMS to perform the supine-to-stand task.

SST ability was assessed in different neurological diseases. SST duration has been measured in children with developmental disorders between 4-7 years old . It has been used to assess frailty in patients with Parkinson's disease . Its validity and reliability have recently been tested in patients with stroke . Considering the balance, falls and coordination complaints of MS patients, there is a need to measure SST ability and investigate it with other clinical tests. In particular, not being able to stand up after falling problems and staying in a supine position causes loss of motivation and decreases in quality of life for patients. In order to prevent this problem in neurological diseases, it is necessary to evaluate and treat it by working functionally as a result of this evaluation. In MS patients, especially as the EDSS level increases, balance problems and walking problems increase and muscle strength decreases. In these cases, problems of transition between positions and movements come to the fore.

Therefore, SST test can be used as a marker to show functional motor competence of MS patients. SST can be a quick and easy measurement tool to evaluate the effectiveness of rehabilitation. The aim of this study was to investigate the reliability and validity of SST in pwMS.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with revised 2017 McDonald criteria,
* aged older than 18 years,
* ability to walk with or without aid,
* no medication changes in the last 2 months,
* volunteering to participate in the research,
* not having any obstacles to verbal and cognitive communication.

Exclusion Criteria:

* having orthopedic, psychological, and other neurological disorders, having had -a relapse in the past 3 months
* having pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PATIENTS DIAGNOSED WITH MULTIPLE SCLEROSIS ADMITTED TO THE NEUROLOGY OUTPATIENT CLINIC OF SANKO UNİVERSİTESİ SANİ KONUKOĞLU APPLICATION AND RESEARCH HOSPITAL
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Supine-to-stand Test (SST) | 1 years
  The test was used to evaluate supine-to-stand ability. The patients were first laid in a supine position without shoes on a soft mat in a quiet laboratory environment. The patient was asked to stand up with the command "start". The duration time was recorded. The average of the tests repeated twice was recorded
Muscle Strength | 1 years
  Ankle dorsi and plantar flexors strength were evaluated with digital hand dynamometer (Commander Muscle Tester, JTech, Midvale, USA). Ankle muscle strength could predictor for walking capacity in neurological disorders . pwMS performed 3-s maximum isometric voluntary contraction of ankle dorsiflexor and plantar flexors with the dynamometer placed anterior and posterior to the head of metatarsal bones, respectively . Ankle dorsiflexors and plantar flexor strength were tested separately, bilaterally and twice in the supine and prone position, respectively. The average of the values was taken and recorded as Newton.
Nine Hole Test | 1 years
  The 9HPT was used to assess the fine manual dexterity of patients. The patient was instructed to insert pegs into the nine empty pegs on the nine-hole board before removing the pegs while sitting position. The test, which it was designed to be completed as rapidly as possible, was administered bilaterally in two trials for each hand. An average time was reported. The patient's manual dexterity degrades with time. The 9HPT is reliable within and between test sessions, discriminates between healthy participants and pwMS with varying levels of upper limb impairment, and has a good convergent validity with other manual dexterity and more comprehensive upper limb tests
Berg Balance Test | 1 years
  It was functional measure of balance commonly used in pwMS. The scale consists of 14 functional activities frequently used in daily life (standing up from sitting, standing without support, sitting without support, sitting from standing, transferring, standing with eyes closed, standing with legs together, reaching forward while standing, picking up an object from the floor, looking back, turning 360 degrees, standing on the healthy side of a chair, standing with one foot in front, and standing on one leg). Activities are scored between 0 and 4. If the individual cannot perform the activity, 0 points are given, and if the individual performs it independently, 4 points are given. Low scores indicate impaired balance. The highest score is 56, with 0-20 points indicating impaired balance, 21-40 points indicating acceptable balance, and 41-56 points indicating good balance
Timed Up and Go (TUG) | 1 years
  Test was used for a measure of functional mobility in pwMS . The test measures speed during many functions such as standing up, walking, turning and sitting. In the test, the individual was asked to get up from the chair he was sitting in, walk 3 meters at a safe and normal speed, turn, walk back and sit on the chair and the time was recorded in seconds. As the score increases, pwMS' fear of falling increases.
Six-Minute Walk Test (6MWT) | 1 years
  The Six-Minute Walk Test was used to assess walking endurance, following the technique reported by Goldman et al . Each participant was asked to walk as securely and quickly as possible for six minutes without running in a 10-meter corridor. The distance they walked for six minutes was recorded. The test was performed twice, and the average was recorded in centimeters. As the score increases, individuals' walking capacity increases.
Activity-specific Balance Confidence Scale (ABC) | 1 years
  ABC scale is used to fear of falling. The ABC scale is a self-reported measure of balance confidence that includes 16 items from daily life (indoors and ourdoors activity). The things were graded from 0 (no confidence) to 100 (full confidence). As the score increases, confidence in the activity increases
Multiple Sclerosis Quality of Life-54 | 1 years
  The test was used to assess the quality of life. It consists of 2 main groups, 12 subgroups and 2 independent items, namely composite physical health (BFS) and composite mental health (BMS). A high score obtained from the scale indicates a high level of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: hakan polat, phd, Principal Investigator — Sanko University
Locations (1):
- SANKO University, Gaziantep, şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
will be decided when the study is completed

REFERENCES:
- [Background] VanSant AF. Age differences in movement patterns used by children to rise from a supine position to erect stance. Phys Ther. 1988 Sep;68(9):1330-9. doi: 10.1093/ptj/68.9.1330. PMID 3420166
- [Background] Ng SSM, Chen P, Chan TCW, Chang CHL, Cheng RHY, Chow KKL, Yeung AFM, Liu TW, Ho LYW, Yeung JWF, Xu RH, Tse MMY. Reliability and validity of the supine-to-stand test in people with stroke. J Rehabil Med. 2023 Sep 18;55:jrm12372. doi: 10.2340/jrm.v55.12372. PMID 37721097